CLINICAL TRIAL: NCT03133156
Title: Exercise Regulation of Human Adipose Tissue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 2016-33; R01DK112283 (NIH)
Record Dates: First submitted 2017-02-22; First posted 2017-04-28 (Actual); Results first posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Healthy; Obese; Diabetes Mellitus, Type 2
Keywords: Exercise; Training; Type 2 Diabetes; Mellitus
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Intervention Model Description: The current research will consist of 2 different exercise training protocols. Subjects will be randomized into each Arm based on screening criteria and compared to the control (Arm 1)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Moderate Intensity Training-Healthy Lean (Experimental): Eligible subjects will undergo a 10-week moderate intensity exercise program.
  Interventions: Other: Exercise Intervention
- Moderate Intensity Training-Healthy Overweight/Obese (Experimental): Eligible subjects will undergo a 10-week moderate intensity exercise program.
  Interventions: Other: Exercise Intervention
- Moderate Intensity Training-Overweight/Obese Type 2 Diabetes (Experimental): Eligible subjects will undergo a 10-week moderate intensity exercise program.
  Interventions: Other: Exercise Intervention
- High Intensity Training-Healthy Lean. (Experimental): Eligible subjects will undergo a 10-week high intensity exercise program
  Interventions: Other: Exercise Intervention

INTERVENTIONS:
Other: Exercise Intervention — 10-Week Aerobic Exercise Training

SUMMARY:
The purpose of this study is to determine whether exercise training leads to changes in the white adipose tissue that are beneficial to the body's regulation of sugar and body weight.

DETAILED DESCRIPTION:
The prevalence of obesity and type 2 diabetes in the United States and worldwide has risen dramatically over the last few decades, resulting in an enormous need for new therapies to treat these conditions. The discovery that beiging of subcutaneous white adipose tissue may increase energy expenditure has led to tremendous interest in beige cells as a potential treatment for diabetes and obesity. An established treatment for type 2 diabetes and obesity is endurance exercise training. Exercise training can improve systemic homeostasis, and although adaptations to skeletal muscle play a critical role in these effects, the underlying mechanisms are not fully understood. Moreover, the contributions of other tissues in these beneficial effects of exercise on metabolism have not been intensively investigated. The study team hypothesizes that exercise training results in fundamental changes to white adipose tissue, including beiging, and these adaptations play an important role in the effects of exercise training to improve metabolic homeostasis.

ELIGIBILITY:
Inclusion Criteria:

* Age: 25-55 years old at the time of screening
* Body mass index (BMI) must be:

  * ≥20 and ≤ 27 kg/m2 for lean subjects
  * ≥25 and ≤ 37 kg/m2 for subjects with type 2 diabetes
  * ≥27 and ≤ 37 kg/m2 for obese/overweight subjects
* HbA1c values:

  * ≤5.7 ± 0.1% for lean and overweight/obese subjects
  * 6.5 ± 0.1% - 9.0 ± 0.1% for subjects with type 2 diabetes

Exclusion Criteria:

* Age <25 and >55 years old
* Type 1 Diabetes
* HbA1c ≥ 9.0%
* Heart or lung disease
* Basal-Bolus Insulin regimen
* Use of beta-blockers or thiazolidinediones
* Acute systemic infection accompanied by fever, body aches, or swollen lymph glands
* BMI ≥ 37 kg/m2
* Current dieting or weight loss efforts
* Current pregnant or breastfeeding
* Known history of HIV/AIDS or certain cancers
* Biochemical evidence of renal or hepatic dysfunction; renal or liver disease
* Demyelinating diseases such as multiple sclerosis or amyotrophic lateral sclerosis
* Recent blood donation
* Clinical history of stroke
* Severe hypertension (systolic > 160 mmHg or diastolic > 90 mmHg)
* Inability to exercise at 50% of predicted heart rate (HR) reserve at baseline
* Participants who screen positive for The American Heart Association's contraindications to exercise testing
* History of keloid formation

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurie J Goodyear, PhD, Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Moderate Intensity Training-Healthy Lean | Moderate Intensity Training-Healthy Overweight/Obese | Moderate Intensity Training-Overweight/Obese Type 2 Diabetes | High Intensity Training-Healthy Lean
Started | 35 | 35 | 11 | 12
Completed | 26 | 28 | 10 | 10
Not Completed | 9 | 7 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Groups included sedentary adults aged 25-55: lean, overweight/obese without T2DM, and overweight/obese with T2DM. Equal numbers of males and females were enrolled where possible. Participants who did not complete baseline assessments were excluded.
Groups:
- Total: Total of all reporting groups
Arm/Group | Moderate Intensity Training-Healthy Lean | Moderate Intensity Training-Healthy Overweight/Obese | Moderate Intensity Training-Overweight/Obese Type 2 Diabetes | High Intensity Training-Healthy Lean. | Total
Number analyzed (Participants) | 35 | 35 | 11 | 12 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (8) | 38.9 (8.5) | 49.6 (5.1) | 36.9 (9.7) | 38.8 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 19 | 8 | 6 | 48
  Male | 20 | 16 | 3 | 6 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 0 | 2 | 11
  Not Hispanic or Latino | 28 | 27 | 10 | 6 | 71
  Unknown or Not Reported | 2 | 4 | 1 | 4 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 10 | 5 | 1 | 4 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 0 | 3
  White | 21 | 28 | 8 | 8 | 65
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 3 | 1 | 0 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 35 | 35 | 11 | 12 | 93
Body Fat Percentage (via Bioelectrical Impedance Analysis [Mean (Standard Deviation); unit: Body Fat %] — Population: "Body fat percentage data unavailable due to recording error."
  Body Fat %
    number analyzed (Participants) | 34 | 35 | 11 | 12 | 92
    (all) | 24.49 (6.65) | 35.04 (7.69) | 38.42 (6.71) | 26.60 (7.71) | 30.44 (9)
Bodyweight [Mean (Standard Deviation); unit: kilograms] | 70.21 (8.81) | 88.04 (11.89) | 83.01 (8.42) | 73.03 (11.19) | 78.8 (13)
Body Fat Mass [Mean (Standard Deviation); unit: kilograms] — Population: Body fat mass data unavailable due to a recording error.
  kilograms
    number analyzed (Participants) | 34 | 35 | 11 | 12 | 92
    (all) | 24.49 (6.65) | 30.75 (7.94) | 32.01 (6.74) | 19.31 (5.38) | 24.4 (9.2)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Human Adipose Tissue Characteristics Following Exercise Training
Description: Body fat percentage measured before and after exercise training with a bioelectrical impedance scale.
Time Frame: Baseline measurement (week 0, prior to starting exercise training) and post-intervention measurement at week 10, after completion of exercise training.
Measure: Mean (Standard Deviation); unit: body fat %
Arm/Group | Moderate Intensity Training-Healthy Lean | Moderate Intensity Training-Healthy Overweight/Obese | Moderate Intensity Training-Overweight/Obese Type 2 Diabetes | High Intensity Training-Healthy Lean
Number analyzed (Participants) | 26 | 28 | 10 | 10
body fat %
  pre-training | 25.45 (6.34) | 34.12 (7.97) | 38.06 (6.96) | 27.05 (7.70)
  post-training | 25.38 (7.02) | 33.90 (8.60) | 37.20 (7.31) | 25.32 (7.57)

2. Primary Outcome: Changes in Human Adipose Tissue Characteristics Following Exercise Training
Description: Body fat mass measured before and after exercise training with a bioelectrical impedance scale.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Moderate Intensity Training-Healthy Lean | Moderate Intensity Training-Healthy Overweight/Obese | Moderate Intensity Training-Overweight/Obese Type 2 Diabetes | High Intensity Training-Healthy Lean
Number analyzed (Participants) | 26 | 28 | 10 | 10
kilograms
  pre-training | 17.83 (4.38) | 29.96 (7.55) | 31.47 (6.85) | 19.76 (5.54)
  post-training | 17.69 (4.72) | 29.61 (8.22) | 30.61 (7.23) | 18.11 (5.81)

3. Primary Outcome: Changes in Human Adipose Tissue Characteristics Following Exercise Training
Description: Body weight measured before and after exercise training with a bioelectrical impedance scale.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Moderate Intensity Training-Healthy Lean | Moderate Intensity Training-Healthy Overweight/Obese | Moderate Intensity Training-Overweight/Obese Type 2 Diabetes | High Intensity Training-Healthy Lean
Number analyzed (Participants) | 26 | 28 | 10 | 10
kilograms
  pre-training | 70.55 (8.99) | 88.22 (10.47) | 82.4 (8.62) | 73.27 (12.07)
  post-training | 70.4 (8.67) | 87.59 (10.8) | 81.90 (8.97) | 71.81 (12.78)

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Moderate Intensity Training-Healthy Lean | Moderate Intensity Training-Healthy Overweight/Obese | Moderate Intensity Training-Overweight/Obese Type 2 Diabetes | High Intensity Training-Healthy Lean
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35 | 0/11 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35 | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 2/35 | 1/35 | 1/11 | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Moderate Intensity Training-Healthy Lean (N=35) | Moderate Intensity Training-Healthy Overweight/Obese (N=35) | Moderate Intensity Training-Overweight/Obese Type 2 Diabetes (N=11) | High Intensity Training-Healthy Lean (N=12)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Knee Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Ankle Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle Cramp (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Parethesia (Nervous system disorders) | 0 | 1 | 0 | 0
Chest Discomfort (Cardiac disorders) | 1 | 0 | 0 | 0
Lightheadedness (Nervous system disorders) | 0 | 0 | 1 | 0
Toe Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-24): https://cdn.clinicaltrials.gov/large-docs/56/NCT03133156/Prot_SAP_000.pdf
  • Informed Consent Form (2023-07-21): https://cdn.clinicaltrials.gov/large-docs/56/NCT03133156/ICF_001.pdf